CLINICAL TRIAL: NCT02538848
Title: A First in Human, Randomized, Double-Blind Study to Assess Safety and Tolerability, Pharmacokinetic and Pharmacodynamic Effects of HTD4010 in Healthy Participants
Brief Title: Study of HTD4010 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HighTide Biopharma Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4010.PCT001
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 50mg in SAD (Experimental): single dose of 50mg HTD4010 or placebo injectable in healthy volunteers
  Interventions: Drug: HTD4010
- 100mg in SAD (Experimental): single dose of 100mg HTD4010 or placebo injectable in healthy volunteers
  Interventions: Drug: HTD4010
- 200mg in SAD (Experimental): single dose of 200mg HTD4010 or placebo injectable in healthy volunteers
  Interventions: Drug: HTD4010
- 300mg in SAD (Experimental): single dose of 300mg HTD4010 or placebo injectable in healthy volunteers
  Interventions: Drug: HTD4010

INTERVENTIONS:
Drug: HTD4010 — injectable solution
  Other Names: analog of INGAP peptide

SUMMARY:
To investigate safety and tolerability of HTD4010 after single ascending doses (SAD) in healthy volunteers

DETAILED DESCRIPTION:
Safety, tolerability and pharmacokinetics(PK) assessments are the outcome measure.

ELIGIBILITY:
For volunteers in SAD:

Inclusion Criteria:

1. Body mass index (BMI) ≥18.0 to ≤ 30.0 kg/m2
2. Non-diabetic, fasting plasma glucose < 5.6 mmol/L
3. Females must be non-pregnant and non-lactating, and either surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or post-menopausal for ≥12 months.

   Males must be surgically sterile, abstinent or if engaged in sexual relations of child-bearing potential, the participant and his partner must be using an acceptable, highly effective, contraceptive method from screening and for a period of 60 days after the last dose of Study Drug.
4. Ability to provide written informed consent.

Exclusion Criteria:

1. Systolic blood pressure >160 mmHg and/or diastolic blood pressure >90 mmHg at screening.
2. Pregnant or lactating women
3. Participation in an investigational study within 30 days prior to dosing or 5 half-lives within the last dose of investigational product whichever is longer.
4. Current use of any prescription or over-the-counter (OTC) medications, including herbal products and supplements, within 14 days prior to Day 1 or 5 half-lives, whichever is longer. Use of ≤2g paracetamol per day is allowed prior to and during the study at Investigator discretion.
5. Any use of non-steroid anti-inflammatory drugs (NSAIDs) within 7 days prior to dosing.
6. History of any major surgery within 6 months prior to Screening
7. History of any serious adverse reaction or hypersensitivity to any of the product components.
8. Use of parenterally administered proteins or antibodies within 12 weeks of screening.

etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Incidence, severity and causality of adverse events | One day in SAD

CONTACTS AND LOCATIONS:
Overall Officials: Janakan Krishnarajah, Doctor, Principal Investigator — Linear Clinical Research Limited
Locations (1):
- Linear Clinical Research Limited, Perth, Australia